CLINICAL TRIAL: NCT05015452
Title: An Observational Follow-up Assessment of Transcatheter Aortic Valve Implantation in Leipzig
Brief Title: The Leipzig TAVI Registry
Status: Recruiting | Type: Observational
Sponsor: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0089
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — Interventional replacement of the aortic valve

SUMMARY:
A single-center registry including all patients treated with TAVI at the Heart Center, Leipzig, Germany

DETAILED DESCRIPTION:
A single-center registry including all patients treated with transcatheter aortic valve implantation (TAVI) at the Heart Center, Leipzig, Germany. Patients undergo a routine clinical and echocardiographic follow-up schedule, including a long-term follow-up plan up to 10 years to assess valve durability.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with TAVI

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers patient population treated with TAVI
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 10 years
  Cardiovascular and not cardiovascular death
  1. identify the current incidence of periprocedural complications.
  2. identification of risk groups
  3. description of the long-term outcome with special attention to the durability of the different prostheses

SECONDARY OUTCOMES:
Structural valve deterioration | Up to 10 years
  Transposthetic mean pressure gradient ≥ 40mmHg and/or ≥20mmHg rise from baseline OR severe intraprosthetic aortic regurgitation

CONTACTS AND LOCATIONS:
Locations (1):
- Herzzentrum Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Wahab M, Kitamura M, Fitzgerald SJ, Dumpies O, Wilde J, Gohmann RF, Majunke N, Gutberlet M, Kiefer P, Noack T, Lurz P, Desch S, Frawley C, Ward K, Borger MA, Holzhey D, Thiele H. Neo-Commissural Alignment Technique for Transcatheter Aortic Valve Replacement Using the ACURATE Neo Valve. Circ Cardiovasc Interv. 2022 Jul;15(7):e011993. doi: 10.1161/CIRCINTERVENTIONS.122.011993. Epub 2022 Jul 1. No abstract available. PMID 35775417